CLINICAL TRIAL: NCT04165785
Title: Efficiency and Changes of Cytokines Expression in Tear After Intense Pulsed Light Treating Evaporated Dry Eye With Demodicosis
Brief Title: Efficiency and Changes of Cytokines Expression in Tear After Intense Pulsed Light Treating Dry Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 198302
Record Dates: First submitted 2019-11-10; First posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Dry Eye Syndromes
Keywords: Optimal pulsed technology intense pulsed light; meibomian gland dysfunction; demodicosis; Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized 1:1 to a study arm and a control arm. Subjects in the study arm will be treated with OPT IPL and meibomian gland expression. Subjects in the control arm will be treated with sham OPT IPL and meibomian gland expression.
Who Masked: Participant
Masking Description: Subjects in the study arm will receive a series of OPT IPL pulses using the M22 IPL handpiece. In subjects of the control arm, the device will be disabled. The subject will feel the lightguide on the skin, will hear clicking sounds, but no light will be actually produced by the M22 device. Since during treatment both eyes of the subject will be fully occluded, no subject will be able to see if the treatment is actual or sham. There is no way to completely mask the subjects, since the IPL generally causes slight redness of the skin, and in some patients is may also cause some discomfort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- OPT IPL followed by MGX (Experimental): Subjects in the experimental arm will receive OPT IPL followed by MGX: OPT IPL pulses will be administered on the skin of the malar region (both cheeks, from tragus to tragus including the nose) and below the lower eyelids. Following OPT IPL therapy, subjects will undergo MGX of both eyelids in both eyes.
  Interventions:
  Device: IPL Procedure: MGX
  Interventions: Device: OPT IPL; Procedure: MGX
- Sham OPT IPL followed by MGX (Sham Comparator): Subjects in the sham comparator arm will receive Sham OPT IPL followed by MGX: Sham OPT IPL pulses will be administered on the skin of the malar region (both cheeks, from tragus to tragus including the nose) and below the lower eyelids. Following Sham OPT IPL therapy, subjects will undergo MGX of both eyelids in both eyes.
  Interventions:
  Device: Sham IPL Procedure: MGX
  Interventions: Device: Sham OPT IPL; Procedure: MGX

INTERVENTIONS:
Device: OPT IPL — Intense pulsed light (IPL) is a non-invasive and non-laser light treatment that is FDA-approved for various conditions in dermatology. Subjects will receive a total of 4 IPL treatments over the course of the study, at intervals of 2 weeks. Each treatment will include applications of 24 IPL pulses in the malar region and close to the lower eyelids, followed by meibomian gland expression.
  Arms: OPT IPL followed by MGX
Device: Sham OPT IPL — Sham Optimal pulsed technology intense pulsed light IPL will be implemented with an IPL device in which all light is blocked by a filter. Subjects will receive a total of 4 sham treatments over the course of the study, at intervals of 2 weeks. Each treatment will include applications of 24 sham pulses in the malar region and close to the lower eyelids, followed by meibomian gland expression.
  Arms: Sham OPT IPL followed by MGX
Procedure: MGX — Meibomian gland expression (MGX) will be implemented by squeezing the meibomian glands with the aid of stainless steel jaeger lid plate positioned in the inferior fornix space between the tarsal and bulbar conjunctiva, and a cotton swab in another side.

SUMMARY:
The aim of the current study is to investigate changes of tear cytokines levels as well as the efficacy and the reduction of demodex infestation after OPT IPL treatment in patients with meibomian gland dysfunction-Associated demodicosis. The effect of OPT IPL will be examined in a study designed as a randomised controlled trial. In the study arm, subjects will undergo 4 treatment sessions, consisting of OPT IPL pulses immediately followed by meibomian gland expression (MGX). In the control arm, subjects will undergo the same treatments, except that the OPT IPL pulses will be disabled. For each subject, the duration of the study will be 2 months , as explained in the detailed description.

DETAILED DESCRIPTION:
All subjects will receive 4 treatments at 2 weeks intervals. In each treatment session, a subject allocated to the study group will be treated with Optimal pulsed technology intense pulsed light (OPT IPL) administered in the malar region, from tragus to tragus including the nose, 2-3 mm below the lower eyelids. Immediately following the OPT IPL administration, the subject will undergo meibomian gland expression (MGX) in both eyelids of both eyes. Subjects in the control arm will receive exactly the same treatment, except that the OPT IPL administration will be sham. A single follow-up will occur at 2 months after the baseline (or 2 weeks after the 4th treatment session). At the follow-up, the changes in the outcome measures will be evaluated, and compared between the two arms.

For each subject, the duration of the study will be 2 months: 1st treatment at baseline; 2nd treatment at 2 weeks after baseline; 3rd treatment at 4 weeks after baseline; 4th treatment at 6 weeks after baseline; and a single follow-up at 8 weeks after baseline).

Statistically significant differences between the two arms will support the study hypothesis that IPL treatment is potentially reduce demodex counts and decrease levels of cytokines , and relief to both signs and symptoms of dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to read, understand and sign an Informed Consent (IC) form
* 18-100 years of age
* Subject is able and willing to comply with the treatment/follow-up (FU) schedule and requirements
* In the study eye, tear break up time ≤ 7 seconds
* In the study eye, Meibomian Gland Score (MGS) ≤ 12
* In the study eye, at least 5 non-atrophied meibomian glands in the lower eyelid
* Symptoms self-assessed using the Ocular Surface Disease Index (OSDI) questionnaire ≥ 23

Exclusion Criteria:

* Fitzpatrick skin type V or VI
* Contact lens wear within the month prior to screening
* Unwilling to discontinue use of contact lenses for the duration of the study
* Ocular surgery or eyelid surgery, within 6 months prior to screening
* Neuro-paralysis in the planned treatment area, within 6 months prior to screening
* Other uncontrolled eye disorders affecting the ocular surface, for example active allergies
* Current use of punctal plugs
* Pre-cancerous lesions, skin cancer or pigmented lesions in the planned treatment area
* Uncontrolled infections or uncontrolled immunosuppressive diseases
* Subjects with ocular infections, within 6 months prior to screening
* Prior history of cold sores or rashes in the perioral area or in the planned treatment area that could be stimulated by light at a wavelength of 560 nm to 1200 nm, including: Herpes simplex 1 & 2, Systemic Lupus erythematosus, and porphyria
* Within 3 months prior to screening, use of photosensitive medication and/or herbs that may cause sensitivity to 560-1200 nm light exposure, including: Isotretinoin, Tetracycline, Doxycycline, and St. John's Wort
* Over exposure to sun, within 4 weeks prior to screening
* Use of prescription eye drops for dry eye, within 7 days prior to screening, excluding artificial tears and glaucoma drops
* Radiation therapy to the head or neck, within 12 months prior to screening
* Planned radiation therapy, within 8 weeks after the last treatment session
* Treatment with chemotherapeutic agent, within 8 weeks prior to screening
* Planned chemotherapy, within 8 weeks after the last treatment session
* New topical treatments within the area to be treated, or oral therapies, within 3 months prior to screening- except over-the-counter acetaminophen-based analgesics for pain management, new oral omega 3 fatty acid supplements and topical artificial tears
* Change in dosage of any systemic medication, within 3 months prior to screening
* Anticipated relocation or extensive travel outside of the local study area preventing compliance with follow-up over the study period
* Legally blind in either eye
* History of migraines, seizures or epilepsy
* Facial IPL treatment, within 12 months prior to screening
* Any thermal treatment of the eyelids, including Lipiflow, within 6 months prior to screening
* Expression of the meibomian glands, within 6 months prior to screening
* In either eye, moderate to severe (Grade 3-4) inflammation of the conjunctiva, including: allergic, vernal or giant papillary conjunctivitis
* In either eye, severe (Grade 4) inflammation of the eyelid, including: blepharochalasis, staphylococcal blepharitis or seborrheic blepharitis
* Ocular surface abnormality that may compromise corneal integrity in either eye (e.g., prior chemical burn, recurrent corneal erosion, corneal epithelial defect, Grade 3 corneal fluorescein staining, or map dot fingerprint dystrophy)
* Eyelid abnormalities that affect lid function in either eye, including: entropion, ectropion, tumor, edema, blepharospasm, lagophthalmos, severe trichiasis, and severe ptosis
* Any systemic condition that may cause dry eye disease, including: Stevens-Johnson syndrome, vitamin A deficiency, rheumatoid arthritis, Wegener's granulomatosis, sarcoidosis, leukemia, Riley-Day syndrome, systemic lupus erythematosus, and Sjögren's syndrome
* Unwilling or unable to abstain from the use of medications known to cause dryness (e.g., isotretinoin, antihistamines) throughout the study duration. Subjects must discontinue these medications for at least 1 month prior to the baseline visit.
* Any condition revealed whereby the investigator deems the subject inappropriate for this study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-07-28 (Actual)

PRIMARY OUTCOMES:
change of baseline demodex counts | 2 months
  Six lashes with cylindrical dandruff (CD) were epilated from each eye (3 in upper eyelid and 3 in lower eyelid) under slit lamp and mounted on glass slides and were examined under optical microscopy to confirm the presence of D folliculorum. Demodex counts greater than or equal to 1 were Demodex-positive.
change of baseline tear cytokines levels | 2 months
  Change of IL-1α, IL-1β, IL-6, IL-7, IL-12p40, IL-13, IL-17A, IL-8, MMP-3, MMP-9 in the study eye, from baseline to follow-up, in both eyes

SECONDARY OUTCOMES:
Change from baseline of Ocular Surface Disease Index score | 2 months
  The ocular surface disease index score was assessed as a subjective parameter to evaluate the ocular symptoms of dry eye on a score of zero to 100, and subject with a score of greater than 12 was considered abnormal.
change from baseline of schirmer I test | 2 months
  Schirmer I test (without anesthesia) was used to assess tear production by inserting in each eye a sterile dry strip (Jingming, Tianjin, China) into the lateral canthus of the lower eyelid away from the cornea over 5 minutes. The length of the strip that was wetted by absorbed tears was then measured in millimeter to evaluate tear secretion function. Values of less than 7.0 mm are considered a diagnosis of aqueous tear deficiency.
change from baseline of the Lid margin abnormalities score | 2 months
  The slit-lamp biomicroscopy was used to score the lid margin abnormalities: the following four parameters were scored as 0 (absent) or 1 (present) of lid margin abnormalities: lid margin irregularity, plugging of the meibomian orifices, lid margin vascular engorgement, and anterior or posterior replacement of mucocutaneous junction. The sum was recorded as 0-4.
change from baseline of meibum grade score | 2 months
  Meibum grade was assessed in each of eight glands of the central third of the lower lid on a scale of zero to three for each gland: zero (clear), one (cloudy), two (cloudy with debris, granular) and three (thick, like toothpaste). Total score range, 0 to 24
change from baseline of corneal fluorescein staining score | 2 months
  The corneal fluorescein staining score was assessed by instilling fluorescein into the lower conjunctival sac with a fluorescein strip (Jingming, Tianjin, China) moistened with preservative-free saline solution. The grading system recommended by NEI divides the cornea into 5 zones (central, superior, temporal, nasal and inferior). For each zone, the corneal fluorescein staining score was graded on a scale from 0 to 3. Therefore, the maximum score was 15
change of baseline of lashes in vivo confocal microscopy laser | 2 months
  In vivo confocal microscopy laser (IVCM, HRTII Cornea Module; Heidelberg Engineering GmbH, Dossenheim, Germany) was used to examine almost 10-20 eyelashes in both eyes. Demodex folliculorum identified in the infundibulum of the eyelashes and the space adjacent to the eyelash shafts as hypo-reflective elongated bodies with a hyperreflective head. Demodex counts greater than or equal to 1were considered positive.
change from baseline of fluorescein tear break up time | 2 months
  The fluorescein tear beak up time was evaluated immediately after the assessment of staining. The patient was required to blink several times to ensure adequate coating of the dye on the cornea. Using a cobalt blue filter and slit-lamp biomicroscopy, the interval between the last complete blink and appearance of the first dry spot in the stained tear film was recorded as the fluorescein tear beak up time. The test was repeated 3 times and the average fluorescein tear beak up time was calculated in second. Values of less than 10 seconds are considered abnormal.

CONTACTS AND LOCATIONS:
Locations (1):
- The First affiliated hospital of harbin medical university, Harbin, Heilongjiang, China

IPD SHARING:
Plan to Share IPD: No